CLINICAL TRIAL: NCT02818790
Title: PREventive Care Infrastructure Based On Ubiquitous Sensing (PRECIOUS)
Brief Title: PREventive Care Infrastructure Based On Ubiquitous Sensing (PRECIOUS). VHIR Pilot.
Acronym: PRECIOUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Aalto University (Other); University of Helsinki (Other); Firstbeat Technologies Ltd. (Industry); University of Vienna (Other); Telecom Bretagne (Unknown); Campden BRI (Unknown); EuroFIR (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRECIOUS_VHIR_Pilot (611366)
Record Dates: First submitted 2016-06-16; First posted 2016-06-30 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Obesity
Keywords: mHealth; Motivational Interviewing; Obesity; Prevention; Diet; Physical Activity; Health Preventive System
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1. Control (No Intervention)
- Group 2. Intervention 1 (Experimental)
  Interventions: Behavioral: Intervention 1
- Group 2. Intervention 2 (Experimental)
  Interventions: Behavioral: Intervention 2

INTERVENTIONS:
Behavioral: Intervention 1 — Bodyguard + Precious App. Short onsite training session on how to use the system.
  Arms: Group 2. Intervention 1
Behavioral: Intervention 2 — Bodyguard + Precious App + Motivational Interviewing. Face to face counseling session followed by a short onsite training session on how to use the system.
  Arms: Group 2. Intervention 2

SUMMARY:
The goal of the MI field test is to assess users' overall satisfaction, usability and acceptability of the PRECIOUS system, and to explore if MI in combination with gamification principles is a feasible solution to foster adherence to PRECIOUS system. Moreover, it is pursued to trigger behavior change and build up motivation to maintain sustained change towards healthy lifestyles. The field test at University Hospital Vall d'Hebron will be carried out with morbidly obese pre-diabetic patients. This pilot test will serve to explore users' acceptance of PRECIOUS system in an early stage of its development. Considering that this is a pilot test, feedback and outcomes obtained will serve to refine and adjust PRECIOUS system concept and architecture.

DETAILED DESCRIPTION:
The pilot test will recruit 30 morbidly obese pre-diabetic patient and they will be randomized into three groups: Group 1. Treatment as usual; Group 2. PRECIOUS system; Group 3. PRECIOUS system and Motivational Interviewing counseling. Researchers of this study will contact telephonically with potential participants and will ask for voluntary participation. Among those who agree, a face-to-face appointment at the reference hospital will be scheduled. In this appointment, general information on the study objectives and procedures will be offered.

The length of intervention will be 3 months with the following scheduled follow-up appointments: week 2 (considering baseline as week 1), week 5, week 8 and week 12. In the follow-up appointments 2, 5 and 8, only doubts and questions regarding system use will be addressed (not specific measures will be collected). Two types of measures will be assessed: 1) Primary outcome measures (at the end of the test) to assess usability, satisfaction, user's acceptance, and effectiveness of PRECIOUS system; and 2) Secondary outcome measures (baseline and final assessment) to assess different aspects of lifestyle and health habits. In addition, all patients will use a device to record heart rate during 3 consecutive days (week 1 and 12).

ELIGIBILITY:
Inclusion Criteria:

* All patients must be under the care of medical specialists who adheres to national guidelines for morbid obesity or pre-diabetic conditions.
* Age older than 18 years.
* Body max index (BMI): ≥ 30 mg/m2.
* Pre-diabetic condition following ADA criteria: fasting plasma glucose level from 5.6mmol/L (100 mg/dL) to 6.9mmol/L (125 mg/dL).
* Patients must be able to participate, understand and complete questionnaires in Spanish language.
* Patients must refer to be used to use multimedia platforms such as PDAs, tablets, laptops, smart phones or personal computers in a regular basis.

Exclusion Criteria:

* Any mental (e.g. cognitive impairment, severe psychopathology not stabilized) or physical condition that could interfere with the successful application of the research protocol.
* Patients will be recruited from specialist outpatient consultation at Vall d'Hebron Research Institute (VHIR). All patients must be under the care of specialists who adhere to national guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Patients' subjective assessment of usability of the PRECIOUS system | At the end of the test (Session 5, week 12)
  o Numeric scale 0-10 & 10 items, 5-point Likert Scale, 0-100
Satisfaction with the PRECIOUS system | At the end of the test (Session 5, week 12)
  o 16 Numeric scales 0-10
User's acceptance of the PRECIOUS system | At the end of the test (Session 5, week 12)
  o 4 Numeric scales 0-10, based on QUIS7
Effectiveness of the PRECIOUS system | At the end of the test (Session 5, week 12)
  o Difference between the control group and the intervention groups regarding engagement and adherence to targeted healthy habits based on MCID between groups of the PRECIOUS system.

SECONDARY OUTCOMES:
Demographics and clinical data | Session 1 (week 1) and Session 5 (week 12)
  o Ad hoc protocol (17 items)
Health-related quality of life | Session 1 (week 1) and Session 5 (week 12)
  o SF12v2: 12 items
Weight management | Session 1 (week 1) and Session 5 (week 12)
  o S-Weight (5 items) & P-Weight (34 items)
Severity of the core symptoms of Depression, Anxiety & Stress | Session 1 (week 1) and Session 5 (week 12)
  o DASS (21 items)
Physical activity | Continuous measure (intervention groups)
  o Data provided by the app
Nutritional habits | Continuous measure (intervention groups)
  o Data provided by the app
Alcohol consumption | Session 1 (week 1) and Session 5 (week 12)
  o Audit (10 items)
Tobacco use | Session 1 (week 1) and Session 5 (week 12)
  o Fagerström (6 items)
Sleep quality | Session 1 (week 1) and Session 5 (week 12)
  o Pittsburg Quality of Sleep index (18 items)
Assessment of the motivational aspects of PRECIOUS | Session 5 (week 12) Intervention groups
  o 23 numeric scales 0-10
Bodyguard 2 device | Session 1 (week 1) and Session 5 (week 12)
  Heart Rate Variability measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jose Costa Requena, PhD, Study Chair — Aalto University; Pilar Lusilla Palacios, PhD, MD, Principal Investigator — Hospital Universitari Vall d'Hebron - Fundació Institut de Recerca Vall d'Hebron. Department of Psychiatry
Locations (1):
- Hospital Universitari Vall d'Hebron - Fundació Institut de Recerca Vall d'Hebron. Department of Psychiatry, Barcelona, Spain

REFERENCES:
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Castellano-Tejedor C, Moreno J, Ciudin A, Parramon G, Lusilla-Palacios P. PREventive Care Infrastructure based On Ubiquitous Sensing (PRECIOUS): A Study Protocol. JMIR Res Protoc. 2017 May 31;6(5):e105. doi: 10.2196/resprot.6973. PMID 28566263
- See also: Link of full list of publications of the consortium of the PRECIOUS Project — http://www.thepreciousproject.eu/?page_id=15